CLINICAL TRIAL: NCT02993250
Title: A Phase 2a, Multicenter, Open-label Study to Investigate the Safety, Pharmacokinetics, and Efficacy of Combination Treatment of AL-335, Odalasvir, and Simeprevir in Japanese Subjects With Chronic Hepatitis C Genotype 1 or 2 Virus Infection, With or Without Compensated Cirrhosis Who Are Direct Acting Antiviral Treatment-naïve
Brief Title: A Study to Investigate the Safety, Pharmacokinetics, and Efficacy of Combination Treatment of AL-335, Odalasvir, and Simeprevir in Japanese Participants With Chronic Hepatitis C Genotype 1 or 2 Virus Infection, With or Without Compensated Cirrhosis Who Are Direct Acting Antiviral Treatment-naive
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Janssen Pharmaceutical K.K. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR108264; 64294178HPC2003 (Other: Janssen Pharmaceutical K.K., Japan)
Record Dates: First submitted 2016-12-13; First posted 2016-12-15 (Estimated); Results first posted 2019-09-11 (Actual); Last update posted 2019-09-11 (Actual); Status verified 2019-09

CONDITIONS: Hepatitis C, Chronic
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — adafosbuvir; odalasvir; Simeprevir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cohort 1 (Chronic Hepatitis C Without Cirrhosis) (Experimental): Participants will receive 800 milligram (mg) AL-335 +odalasvir (ODV) 25 mg+simeprevir (SMV) 75 mg once daily for 8 weeks in Cohort 1.
  Interventions: Drug: AL-335; Drug: Odalasvir (ODV); Drug: Simeprevir (SMV)
- Cohort 2 (Chronic Hepatitis C With Compensated Cirrhosis) (Experimental): Participants will receive AL-335 800 milligram (mg)+ODV 25 mg+SMV 75 mg once daily for 12 weeks in Cohort 2. Dosing in cohort 2 will be started according to decision of Data Review Committee (DRC).
  Interventions: Drug: AL-335; Drug: Odalasvir (ODV); Drug: Simeprevir (SMV)

INTERVENTIONS:
Drug: AL-335 — Participants will receive AL-335 800 mg once daily for 8 weeks in cohort 1 and 12 weeks in cohort 2.
  Other Names: JNJ-64146212
Drug: Odalasvir (ODV) — Participants will receive ODV 25 mg once daily for 8 weeks in cohort 1 and 12 weeks in cohort 2.
  Other Names: JNJ-64289901
Drug: Simeprevir (SMV) — Participants will receive SMV 75 mg once daily for 8 weeks in cohort 1 and 12 weeks in cohort 2.
  Other Names: TMC435

SUMMARY:
The main purpose of this study is to evaluate the safety and tolerability of a combination treatment of AL-335, odalasvir (ODV), and simeprevir (SMV) for 8 weeks in Japanese participants with genotype 1 or 2 chronic hepatitis C virus (HCV) infection without cirrhosis and for 12 weeks in direct-acting antiviral (DAA)-naive Japanese participants with genotype 1 or 2 chronic HCV infection with compensated cirrhosis.

ELIGIBILITY:
Inclusion Criteria:

* Chronic hepatitis C virus (HCV) infection
* All participants must have HCV genotype 1 or 2 infection, determined at screening
* HCV ribonucleic acid (RNA) plasma levels greater than or equal to (>=)10,000 international units per Milliliter (IU/mL), determined at screening
* Direct-acting antiviral (DAA)-naive participants, defined as not having received treatment with any approved or investigational DAA drug for chronic HCV infection; prior HCV therapy consisting of interferon (IFN, pegylated or nonpegylated) with or without ribavirin (RBV) is allowed
* Participants without cirrhosis or with compensated cirrhosis

Exclusion Criteria:

* Infection with HCV genotype - 3, 4, 5, or 6
* Co-infection with human immunodeficiency virus (HIV 1 or HIV 2 antibody positive) or hepatitis B virus (HBV) (hepatitis B surface antigen [HBsAg] positive)
* Prior treatment with any investigational or approved HCV DAA, either in combination with PegIFN or IFN free
* Any evidence of liver disease of non-HCV etiology. This includes, but is not limited to, acute hepatitis A infection (immunoglobulin M), drug or alcohol related liver disease, autoimmune hepatitis, hemochromatosis, Wilson's disease, alpha 1 antitrypsin deficiency, primary biliary cirrhosis, or any other non-HCV liver disease that is considered clinically significant by the investigator
* Evidence of hepatic decompensation as assessed with Child-Pugh Class B or C or any of the following: history or current clinical evidence of ascites, bleeding varices, or hepatic encephalopathy

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2016-12-21 (Actual); Primary Completion 2018-05-07 (Actual); Study Completion 2018-05-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Pharmaceutical K.K., Japan Clinical Trial, Study Director — Janssen Pharmaceutical K.K.
Locations (14):
- Japan (14):
  - Amagasaki-shi
  - Bunkyō City
  - Hiroshima
  - Kagoshima
  - Kurume-shi
  - Musashino-shi
  - Nagoya
  - Omura-shi
  - Osaka
  - Saitama
  - Sakaishi
  - Sapporo
  - Suita-shi
  - Yokohama

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort 1: Chronic Hepatitis C Without Cirrhosis: Participants received AL-335 800 milligram (mg) (2*400) tablets, odalasvir (ODV) 25 mg tablet and simeprevir (SMV) 75 mg capsule once daily orally for 8 weeks.
- Cohort 2: Chronic Hepatitis C With Compensated Cirrhosis: Participants received AL-335 800 mg (2*400) tablets, ODV 25 mg tablet and SMV 75 mg capsule once daily orally for 12 weeks.
Period: Overall Study
Arm/Group | Cohort 1: Chronic Hepatitis C Without Cirrhosis | Cohort 2: Chronic Hepatitis C With Compensated Cirrhosis
Started | 22 | 11
Completed | 22 | 10
Not Completed | 0 | 1
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1: Chronic Hepatitis C Without Cirrhosis | Cohort 2: Chronic Hepatitis C With Compensated Cirrhosis | Total
Number analyzed (Participants) | 22 | 11 | 33
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.3 (11.1) | 54.9 (6.76) | 57.8 (9.98)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 4 | 21
  Male | 5 | 7 | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 22 | 11 | 33
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 22 | 11 | 33
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Japan | 22 | 11 | 33

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events (AEs)
Description: An adverse event was any untoward medical event that occurs in a participant administered an investigational product, and it does not necessarily indicate only events with clear causal relationship with the relevant investigational product.
Time Frame: Approximately 38 weeks (Cohort 1) and 42 weeks (Cohort 2)
Population: The safety analysis set included all enrolled participants who received at least 1 dose of study drug.
Measure: Number; unit: participants
Arm/Group | Cohort 1: Chronic Hepatitis C Without Cirrhosis | Cohort 2: Chronic Hepatitis C With Compensated Cirrhosis
Number analyzed (Participants) | 22 | 11
participants | 15 | 9

2. Secondary Outcome: Percentage of Participants With Sustained Virologic Response 4 Weeks (SVR4) After Actual End-of-Treatment
Description: SVR4 was defined as hepatitis C virus (HCV) ribonucleic acid (RNA) less than (<) lower limit of quantification (LLOQ; 15 international unit per milliliter [IU/mL]) detected or not detected at 4 weeks after the actual End-of-treatment (EOT).
Time Frame: Week 4 (follow-up phase)
Population: Full analysis set included all enrolled participants who received at least 1 dose of study drug (that is AL-335, ODV or SMV) and had at least 1 postbaseline efficacy measurement in this study.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Cohort 1: Chronic Hepatitis C Without Cirrhosis | Cohort 2: Chronic Hepatitis C With Compensated Cirrhosis
Number analyzed (Participants) | 22 | 11
Percentage of participants | 100 [84.6 to 100] | 100 [71.5 to 100]

3. Secondary Outcome: Percentage of Participants With Sustained Virologic Response 12 Weeks (SVR12) After Actual End-of-treatment
Description: SVR12 was defined as HCV RNA < LLOQ (15 IU/mL) detected or not detected at 12 weeks after the actual EOT.
Time Frame: Week 12 (follow-up phase)
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Cohort 1: Chronic Hepatitis C Without Cirrhosis | Cohort 2: Chronic Hepatitis C With Compensated Cirrhosis
Number analyzed (Participants) | 22 | 11
Percentage of participants | 100 [84.6 to 100] | 100 [71.5 to 100]

4. Secondary Outcome: Percentage of Participants With Sustained Virologic Response 24 Weeks (SVR24) After Actual End-of-treatment
Description: SVR 24 was defined as HCV RNA < LLOQ (15 IU/mL) detected or not detected at 24 weeks after the actual EOT.
Time Frame: Week 24 (follow-up phase)
Population: Full analysis set included all enrolled participants who received at least 1 dose of study drug (that is AL-335, ODV or SMV) and had at least 1 postbaseline efficacy measurement in this study. Here, 'N' (number of participants analyzed) signifies those participants who were evaluable for this outcome measure.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Cohort 1: Chronic Hepatitis C Without Cirrhosis | Cohort 2: Chronic Hepatitis C With Compensated Cirrhosis
Number analyzed (Participants) | 22 | 10
Percentage of participants | 100 [84.6 to 100] | 90.9 [58.7 to 99.8]

5. Secondary Outcome: Percentage of Participants With Viral Relapse
Description: Viral relapse was defined as participants who did not achieve SVR12, with HCV RNA < LLOQ (15 IU/mL) at the EOT and confirmed HCV RNA greater than or equal to (>=) LLOQ during follow-up.
Time Frame: End of treatment up to Week 24 (follow up phase)
Population: Full analysis set included all enrolled participants who received at least 1 dose of study drug (that is AL-335, Odalasvir (ODV) or Simeprevir (SMV)] and had at least 1 postbaseline efficacy measurement in this study.
Measure: Number; unit: Percentage of participants
Arm/Group | Cohort 1: Chronic Hepatitis C Without Cirrhosis | Cohort 2: Chronic Hepatitis C With Compensated Cirrhosis
Number analyzed (Participants) | 22 | 11
Percentage of participants | 0 | 0

6. Secondary Outcome: Percentage of Participants With On-treatment Failure
Description: On-treatment failure was defined as participants who did not achieve SVR12, with confirmed HCV RNA >= LLOQ (15 IU/mL) at the actual EOT.
Time Frame: EOT up to Week 12 (follow up phase)
Population: as for outcome 2
Measure: Number; unit: Percentage of Participants
Arm/Group | Cohort 1: Chronic Hepatitis C Without Cirrhosis | Cohort 2: Chronic Hepatitis C With Compensated Cirrhosis
Number analyzed (Participants) | 22 | 11
Percentage of Participants | 0 | 0

7. Secondary Outcome: Percentage of Participants With On-treatment Virologic Response
Description: Percentage of participants with On-treatment Virologic Response with HCV RNA < LLOQ (15 IU/mL), not detected at specified time points during treatment were reported.
Time Frame: Day 2, Day 3, Week 1, 2, 3, 4, 6, 8 (for Cohort 1), 10, and 12 (for Cohort 2 only)
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | Cohort 1: Chronic Hepatitis C Without Cirrhosis | Cohort 2: Chronic Hepatitis C With Compensated Cirrhosis
Number analyzed (Participants) | 22 | 11
Percentage of participants
  Day 2: < 15 IU/mL not detected | 4.5 | 0
  Day 3: < 15 IU/mL not detected | 4.5 | 0
  Week 1: < 15 IU/mL not detected | 4.5 | 18.2
  Week 2: < 15 IU/mL not detected | 22.7 | 45.5
  Week 3: < 15 IU/mL not detected | 54.5 | 63.6
  week 4: < 15 IU/mL not detected | 72.7 | 72.7
  Week 6: < 15 IU/mL not detected | 90.9 | 100
  Week 8: < 15 IU/mL not detected | 100 | 100
  Week 10: < 15 IU/mL not detected: number analyzed (Participants) | 0 | 11
  Week 10: < 15 IU/mL not detected |  | 100
  Week 12: < 15 IU/mL not detected: number analyzed (Participants) | 0 | 11
  Week 12: < 15 IU/mL not detected |  | 100

8. Secondary Outcome: Time to Achieve HCV RNA Not Detected or HCV RNA <LLOQ
Description: Time to Achieve HCV RNA not Detected or HCV RNA <LLOQ (15 IU/mL) was reported.
Time Frame: EOT up to Week 24 (follow up phase)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Cohort 1: Chronic Hepatitis C Without Cirrhosis | Cohort 2: Chronic Hepatitis C With Compensated Cirrhosis
Number analyzed (Participants) | 22 | 11
Days | 19.0 (1.68) | 18.6 (3.86)

ADVERSE EVENTS:
Time Frame: Approximately 38 weeks (Cohort 1) and 42 weeks (Cohort 2)
Description: Safety analysis set included all enrolled participants who received at least 1 dose of study drug (that is AL-335, Odalasvir (ODV) or Simeprevir (SMV)].
Arm/Group | Cohort 1: Chronic Hepatitis C Without Cirrhosis | Cohort 2: Chronic Hepatitis C With Compensated Cirrhosis
All-Cause Mortality (participants affected / at risk) | 0/22 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/22 | 1/11
Other Adverse Events (participants affected / at risk) | 15/22 | 9/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1: Chronic Hepatitis C Without Cirrhosis (N=22) | Cohort 2: Chronic Hepatitis C With Compensated Cirrhosis (N=11)
Cataract (Eye disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1: Chronic Hepatitis C Without Cirrhosis (N=22) | Cohort 2: Chronic Hepatitis C With Compensated Cirrhosis (N=11)
Atrioventricular Block First Degree (Cardiac disorders) | 2 | 1
Supraventricular Extrasystoles (Cardiac disorders) | 0 | 1
Cataract (Eye disorders) | 0 | 1
Eye Discharge (Eye disorders) | 0 | 1
Abdominal Pain Upper (Gastrointestinal disorders) | 2 | 0
Diarrhoea (Gastrointestinal disorders) | 3 | 0
Gastritis (Gastrointestinal disorders) | 0 | 2
Gastrointestinal Motility Disorder (Gastrointestinal disorders) | 0 | 1
Malaise (General disorders) | 2 | 0
Nasopharyngitis (Infections and infestations) | 0 | 1
Oral Herpes (Infections and infestations) | 0 | 1
Viral Upper Respiratory Tract Infection (Infections and infestations) | 1 | 4
Alanine Aminotransferase Increased (Investigations) | 2 | 2
Aspartate Aminotransferase Increased (Investigations) | 2 | 2
Blood Cholesterol Increased (Investigations) | 0 | 1
Neck Pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 0 | 1
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 0 | 1
Headache (Nervous system disorders) | 3 | 2
Eczema (Skin and subcutaneous tissue disorders) | 0 | 1

LIMITATIONS AND CAVEATS:
As the sponsor decided to discontinue the development of JNJ-64294178, the study enrollment to reach the target number of participants was not completed in Cohort 2.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If an investigator wishes to publish information from the study, a copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested by the sponsor in writing, the investigator will withhold such publication for up to an additional 60 days.

DOCUMENTS (2):
  • Statistical Analysis Plan (2018-06-08): https://cdn.clinicaltrials.gov/large-docs/50/NCT02993250/SAP_000.pdf
  • Study Protocol (2017-07-27): https://cdn.clinicaltrials.gov/large-docs/50/NCT02993250/Prot_001.pdf